CLINICAL TRIAL: NCT01975402
Title: Evaluation of the BodyGuardian End-to-end Remote Monitoring Platform in an Outpatient Heart Failure Population
Acronym: R01-Aim2
Status: Completed | Type: Observational
Sponsor: Mayo Clinic (Other)
Collaborators: Preventice (Industry); National Institute on Aging (NIA) (NIH)
Responsible Party: Principal Investigator, Lyle J. Olson, M.D., PI, Mayo Clinic
Other Study IDs: 13-005607; R01AG041676 (NIH)
Record Dates: First submitted 2013-10-23; First posted 2013-11-04 (Estimated); Last update posted 2019-05-21 (Actual); Status verified 2019-05

CONDITIONS: Congestive Heart Failure
Keywords: Congestive Heart Failure
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
We will evaluate the end to end remote monitoring system in a less controlled environment and concurrently develop the infrastructure to support the back end of the system

DETAILED DESCRIPTION:
The overall objective of our research is to test, adapt, refine and validate the BodyGuardian technology and related end-to-end remote monitoring system to be used outside usual medical care environments to reduce hospital readmissions and facilitate independent living for heart failure patients. An important component of our overall strategy for continued development and refinement of the remote monitoring system is the incorporation of iterative behavioral evaluations to facilitate assessment and refinement in order to optimize adherence, utilization, and usability for patients as well as efficiency and functionality for providers.

ELIGIBILITY:
Inclusion Criteria:

* Outpatients
* Stable New York Heart Association Class I-III HF (defined as no admissions for > 1 year)
* Recruited from the Mayo Heart Failure Clinic, including 15 men and 15 women
* Age > 50 years
* Reside in Olmsted County

Exclusion Criteria:

* Hospital admission for HF within past year
* Dementia
* Overall life expectancy < 2 months
* Blindness
* Pregnancy or women able to become pregnant
* Skin allergy to adhesives
* Inadequate cell phone coverage (international patients or international travel during study period)
* Documented Ejection Fraction of >40%

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Individuals >50 years with Congestive Heart Failure
Sampling Method: Probability Sample
Enrollment: 42 (Actual)
Dates: Start 2013-11; Primary Completion 2019-03-31 (Actual); Study Completion 2019-03-31 (Actual)

PRIMARY OUTCOMES:
adherence and utilization of end-to-end system in 30 subjects with stable New York Heart Association class I-III Heart Failure for 2 weeks | 12 months
  To evaluate subject adherence, data transfer, clinical utilization and work-flow as well as perceptions and experiences of HF outpatients (n=30) and providers of the end-to-end remote monitoring system.

SECONDARY OUTCOMES:
effect of end-to-end system on life quality | 12 months
  Evaluation of end-to-end remote monitoring system in a less controlled environment by evaluating ease of use and clinical management.

OTHER OUTCOMES:
Healthcare record integration | 12 months
  Concurrently develop the infrastructure to support the back-end solution of the system including technician support, closed feedback loops to support care of the monitored subjects by an integrated team of health care providers, user-interfaces which display summarized data for the patient and other members of the healthcare team, and integration of summarized data into the Mayo electronic medical record.

CONTACTS AND LOCATIONS:
Overall Officials: Lyle J Olson, MD, Principal Investigator — Mayo Clinic
Locations (3):
- United States (3):
  - Mayo Clinic, Jacksonville, Florida
  - Mayo Clinic Health System-Eau Claire Hospital, Inc., Eau Claire, Wisconsin
  - Mayo Clinic Health System-Franciscan Medical Center, La Crosse, Wisconsin

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials